CLINICAL TRIAL: NCT05616390
Title: A Study to Evaluate the Efficacy and Safety of the Sintilimab Combined With Bevacizumab and Liver Protective Support Therapy in Child-Pugh B and/or ECOG PS 2 Unresectable Hepatocellular Carcinoma
Brief Title: Sintilimab Combined With Bevacizumab and Liver Protective Support Therapy in Unresectable Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L20220940
Record Dates: First submitted 2022-11-08; First posted 2022-11-15 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2022-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Sintilimab; Bevacizumab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — sintilimab; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Sintilimab Combined With Bevacizumab and Liver Protective Support Therapy
  Interventions: Drug: Sintilimab; Drug: Bevacizumab; Combination Product: Liver Protective Support Therapy

INTERVENTIONS:
Drug: Sintilimab — 200mg IV d1,Q3W
  Other Names: IBI308
Drug: Bevacizumab — 7.5mg/kg IV d1,Q3W
Combination Product: Liver Protective Support Therapy — Medical treatment such as liver protection therapy, antiviral therapy, platelet and granulocyte upgrading therapy

SUMMARY:
To evaluate the efficacy and safety of sintilimab combined with bevacizumab and liver protective support therapy in Child-Pugh B and/or ECOG PS 2 unresectable hepatocellular carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Advanced unresectable hepatocellular carcinoma confirmed by histology or cytology
* Age 20-79
* At least one measurable lesion defined in RECIST version 1.1
* Child Pugh grade B
* ECOG PS score 2
* The expected life is at least 90 days

Exclusion Criteria:

* Previously received anti-PD-1, PD-L1, PD-L2, CD137, CTLA-4 antibody treatment, or any other treatment that regulates T cells
* Received systemic corticosteroid or immunosuppressive therapy within 28 days before enrollment
* Complicated with autoimmune diseases or having a history of chronic or recurrent autoimmune diseases
* History of pleural or pericardial adhesions within 28 days before enrollment
* HIV antibody, HTV-Ⅰantibody, HCV antibody, hepatitis B surface protein antigen, hepatitis B surface protein antibody, hepatitis B core protein antibody or any detectable hepatitis B virus DNA test results were positive
* Multiple primary cancers (excluding completely resected basal cell carcinoma, stage I squamous cell carcinoma, carcinoma in situ, intramucosal carcinoma, superficial bladder cancer, and any other cancer that has not recurred for at least 5 years)
* Brain or meningeal metastasis (unless asymptomatic and does not require treatment)
* Uncontrollable or serious cardiovascular disease.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Up to 3 years
  Defined as the proportion of patients with AE, treatment-related AE (TRAE), immune-related AE (irAE), serious adverse event (SAE), assessed by NCI CTCAE v5.0
Overall survival (OS) | Up to 3 years
  Defined as the time from the date of treatment start to the date of death

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 1 years
  Defined as proportion of patients who have a best response of CR or PR
Disease control rate (DCR) | Up to 1 years
  Defined as proportion of patients who have a best response of CR, PR or SD
Quality of Life (QoL) | Up to 3 years
  The improvement in quality of life as measured by the EORTC Quality of Life Questionnaire QLQ-C30 (V3.0)

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China